# CLINICAL TRIAL PROTOCOL: SDP-4-CS202

**Study Title:** A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-Controlled,

Parallel-Group, Study of SDP-4 Ophthalmic Solution in Subjects with Dry Eye

Disease (DED)

**Study Number:** SDP-4-CS202

Study Phase: 2

**Product Name:** SDP-4 Ophthalmic Solution

Indication: Dry eye disease Investigators: Multicenter

**Sponsor:** SilkTech Biopharmaceuticals (SilkTech)

3700 Annapolis Ln. N., Suite 105

Plymouth, MN 55447 Phone: 763-316-4107 Fax: 763-205-5023

**Sponsor Contact:** Brian Lawrence, Ph.D. **Medical Monitor:** Brian Levy, O.D., M.Sc.

3700 Annapolis Ln. N., Suite 105

Plymouth, MN 55447 Phone: 585-978-1943

Email: Safety@Silk-Tech.com

| | Date |
|--------------------|---------------|
| Original Protocol: | 06 March 2020 |

### Confidentiality Statement

The information contained in this document is confidential and proprietary property of Silk Technologies, Ltd. Neither this document nor the information contained herein may be divulged, transmitted, reproduced, published, or otherwise used by others without the express written permission of Silk Technologies, Ltd.

### **SYNOPSIS**

**Sponsor:** SilkTech Biopharmaceuticals

Name of Finished Product: SDP-4 Ophthalmic Solution

Name of Active Ingredient: Silk-Derived Protein-4 (SDP-4; amlisimod)

**Study Title:** 

A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group, Dose-Response Study of SDP-4 Ophthalmic Solution in Subjects with Dry Eye Disease (DED)

Study Number: SDP-4-CS202

Study Phase: 2

### **Primary Objective:**

Assess the safety and efficacy of SDP-4 ophthalmic solution in subjects with DED over an 8-week (56-day) treatment period.

## **Study Design:**

This is a Phase 2, multicenter, double-masked, randomized, vehicle-controlled, parallel-group study designed to evaluate the safety and efficacy of SDP-4 ophthalmic solution in subjects with DED in both eyes (OU) over an 8 week (56-day) treatment period.

Subjects will be randomized to 1.0% SDP-4 Ophthalmic Solution or vehicle in a 1:1 ratio in parallel groups. All investigational products (1.0% SDP-4 and vehicle) will be provided in single-use doses (SUDs) contained in foil pouches. Subjects, the Investigator, and all site personnel responsible for performing study assessments will remain masked to treatment assignment.

Investigational product (IP) will be administered via topical ocular instillation, one drop per eye, twice daily (BID) for 8 weeks (56 days). Both eyes will be treated. A 2-week screening/run-in period on BID vehicle will precede the 8-week randomized treatment period.

Subjects must have a Symptom Assessment in Dry Eye (SANDE) total score of  $\geq$  40 and  $\leq$  70 at Visit 1/Screening and Visit 2/Day 1 to enter the trial. For subjects with a qualifying SANDE score who meet all other inclusion/exclusion criteria, the eye with the lower tear break-up time (TBUT) at Visit 2/Day 1 will be designated as the study eye. In the event both eyes have the same TBUT scores, the eye with the lower Schirmer's test score at Visit 1 will be designated as the study eye. If both eyes have the same TBUT and Schirmer's test scores, the right eye will be designated as the study eye.

The study will consist of 5 clinic visits, 2 visits during the screening/run-in period and 3 on-treatment visits: Visit 1 (Day -14  $\pm$  2/Screening Visit), followed by the 2-week run-in on BID vehicle, Visit 2 (Day 1/Confirmatory and Baseline/Randomization Visit), Visit 3 (Day 14  $\pm$  2), Visit 4 (Day 28  $\pm$  2), and Visit 5 (Day 56  $\pm$  4/End of Study Assessments).

#### **Study Population:**

#### **Number of Subjects Planned:**

A total of 140 randomized subjects are planned, with 70 subjects randomly assigned to each treatment group (1.0% SDP-4 Ophthalmic Solution or vehicle).

#### **Inclusion Criteria:**

Individuals must meet the following criteria at Screening (Visit 1/Day -14) and/or Visit 2/Day 1:

- 1. Willing and able to understand and sign an informed consent form prior to any study-related procedures.
- 2. Male or female patients 18 years of age or older.
- 3. Willing and able to follow study instructions, able to self-administer IP or have IP administered by a caregiver throughout the study period, and able to be present for the required study visits/assessments for the duration of the study.
- 4. Have DED in both eyes, as supported by a subject-reported history of daily symptoms of dry eye for  $\geq 6$  months prior to Visit 1/Screening requiring the use of artificial tears.
- 5. Total score  $\geq$  40 and  $\leq$  70 on the SANDE questionnaire at Visits 1 and 2.
- 6. Tear break-up time (TBUT) of  $\leq$  6 seconds in both eyes at Visits 1 and 2.
- 7. Anesthetized Schirmer's test tear volume  $\geq 3$  mm and <10 mm in both eyes (only at Visit 1).
- 8. Best-corrected visual acuity (BCVA) of +0.7 logMAR or better in each eye as assessed by logMAR chart at Visits 1 and 2.
- 9. Female patients must be 1 year postmenopausal, surgically sterilized, or of childbearing potential with a negative urine pregnancy test at Visit 1/Screening. Females of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include the use of at least one of the following: intrauterine device (IUD), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.

#### **Exclusion Criteria:**

#### Ocular

- 1. Ocular surface corneal disease other than DED.
- 2. Diagnosis of Sjögren's disease.
- 3. Lid margin disorder other than meibomian gland dysfunction (MGD) (e.g., active anterior blepharitis including staphylococcal, demodex or seborrheic; excessive lid laxity, floppy eyelid syndrome, ectropion, entropion) that in the Investigator's opinion could affect study parameters/assessments.
- 4. Presence of any ocular condition (e.g., pterygium) that in the Investigator's opinion could affect study parameters.
- 5. Any previous reconstructive or cosmetic eyelid surgery (e.g., blepharoplasty, ptosis repair, entropion/ectropion repair).
- 6. Any previous invasive glaucoma (e.g., trabeculectomy, shunt) and/or corneal surgery (e.g., penetrating keratoplasty, lamellar keratoplasty, Descemet's stripping endothelial keratoplasty [DSEK]).
- 7. Corneal refractive surgery (e.g., laser-assisted in situ keratomileusis [LASIK], photorefractive keratectomy [PRK], limbal relaxing incision [LRI]) within 12 months prior to Visit 1/Screening.
- 8. Cataract extraction, with or without minimally invasive glaucoma surgery (MIGS) or Yag capsulotomy, within 90 days prior to Visit 1/Screening.
- 9. Cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal within 30 days prior to Visit 1/Screening or planned during the study. If a subject has a punctal plug at Visit 1/Screening for ≥ 30 days and it falls out during the study, it should be replaced with a new plug of the same type.

10. Contact lens wear.

#### **Prior Medications**

- 11. Use of opioids within 90 days prior to Visit 1/Screening.
- 12. Use of isotretinoin (Accutane®) within 60 days prior to Visit 1/Screening.
- 13. Use of topical cyclosporine (Restasis<sup>®</sup>, Cequa<sup>®</sup>) or topical lifitegrast (Xiidra<sup>®</sup>) within 45 days prior to Visit 1/Screening.
- 14. Use of Visine® within 7 days prior to Visit 1/Screening.
- 15. Use of lid scrubs containing chemicals or baby shampoo within 14 days prior to Visit 1/Screening and throughout the study.
- 16. Use of any of the following medications within 30 days prior to Visit 1/Screening and throughout the study:
  - Topical ophthalmic corticosteroids or topical ophthalmic non-steroidal anti-inflammatory drugs (NSAIDs)
  - Autologous serum
  - Topical ophthalmic antibiotics or antivirals
  - Topical ophthalmic antihistamines or mast cell stabilizers
  - Topical ophthalmic medications for lowering of intraocular pressure (IOP) for treatment of glaucoma or ocular hypertension
  - Systemic immunosuppressive agents
  - Systemic (i.e., oral, intravenous, intra-articular, intrathecal, epidural, or intramuscular) corticosteroids (dermatologic steroids other than around the eye or lid are allowed)
  - Tetracycline compounds (tetracycline, doxycycline or minocycline) and systemic cyclosporine

#### **Current Medications**

- 17. Any changes in the dosing of any chronically used systemic drug within 90 days prior to Visit 1/Screening and throughout the study period, including but not limited to the following (if a subject is using an Antihistamine as needed [PRN], it must not be used within 7 days prior to Visit 1/Screening and discontinued throughout the study period):
  - Anticholinergics
  - Antidepressants including selective serotonin reuptake inhibitors (SSRIs), selective serotonin norepinephrine reuptake inhibitors (SSNRIs), tricyclics, and benzodiazepines
  - Antihistamines
  - Systemic H1-receptor antagonists
  - β-adrenoceptor antagonists
  - Calcium channel blockers
- 18. Any changes in the dosing of aspirin and aspirin-containing products within 30 days prior to Visit 1/Screening and throughout the study period.

### **Exclusion Criteria (continued):**

#### General

- 19. Stevens-Johnson syndrome.
- 20. History of immunodeficiency disorder, HIV, positive hepatitis B, C, or evidence of acute active hepatitis A (anti–HAV IgM).
- 21. History of organ or bone marrow transplant.
- 22. History of graft versus host disease (GvHD).
- 23. Systemic lupus erythematosus.
- 24. Chronic pain syndrome (e.g., fibromyalgia).
- 25. Systemic signs of infection (e.g., fever or current treatment with antibiotics).
- 26. Serious systemic disease or uncontrolled medical condition that in the judgment of the Investigator could confound study assessments or limit compliance, including, but not limited to, severe cardiopulmonary disease, uncontrolled hypertension, and/or uncontrolled diabetes.
- 27. Known history of alcohol and/or drug abuse within 12 months prior to Visit 1/Screening that, in the opinion of the Investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject.
- 28. Known allergy or contraindication to any component of IP formulation or diagnostic agents.
- 29. Participation in any drug or device clinical investigation within 30 days prior to Visit 1/Screening and/or during the period of study participation.
- 30. Screening and enrollment of more than one individual who resides in the same household at the same time.
- 31. Screening and enrollment of employees of the clinical site.
- 32. Screening and enrollment of subjects who participated in the SDP-4-CS201 trial.

### **Investigational Product, Dose, and Mode of Administration:**

SDP-4 Ophthalmic Solution (1.0%) 1 drop in each eye BID

### Reference Therapy, Dosage and Mode of Administration:

Vehicle, 1 drop in each eye BID

### **Duration of Treatment:**

Eight (8) weeks (56 days)

#### **Efficacy Assessments:**

- SANDE: Rating on visual analogue scale (0-100 mm) of severity and frequency of dry eye
- Rating on visual analogue scale (0-100 mm) of individual symptoms:
  - Itching
  - Foreign body sensation
  - Burning/stinging
  - Fluctuating vision
  - Eye dryness
  - Eye discomfort
  - Photophobia
  - Eye pain

#### Signs

- TBUT
- Corneal fluorescein staining
- Conjunctival hyperemia

#### **Safety Assessments:**

- Ocular and non-ocular adverse event (AE) monitoring
- BCVA
- Biomicroscopy
- IP comfort assessment

#### **Criteria for Evaluation:**

### **Primary Efficacy Endpoint**

• Mean change from baseline in total SANDE score at Visit 5/Day 56

# **Secondary Efficacy Endpoints**

- Mean and mean change from baseline at each visit for each of the following evaluations:
  - Corneal fluorescein staining (combined and each zone)
  - TBUT
  - Conjunctival hyperemia
  - Individual symptom VAS scores, separately for each symptom
- SANDE
  - Mean change from baseline in total SANDE score at each visit
  - Mean total SANDE score at each visit
  - Mean and mean change from baseline in each component of SANDE at each visit

#### **Statistical Methods:**

A detailed Statistical Analysis Plan (SAP) will be finalized prior to database lock.

#### **General Considerations**

All continuous study assessments will be summarized by treatment and visit (as applicable) using descriptive statistics (n, mean, median, standard deviation, minimum, and maximum). All categorical study assessments will be summarized by treatment and visit (as applicable) using frequency counts and percentages.

All study data will be listed by treatment, subject, and visit (as applicable).

The unit of analysis for efficacy will be the study eye.

## Sample Size Rationale

Based on results from Study SDP-4-CS201, a treatment difference of 12.2 units SANDE total score mean change from baseline at Day 56 was observed in the subgroup population meeting the Total SANDE score  $\geq$  40 and  $\leq$  70. A sample size of 70 subjects per treatment group will have 84.5% power to detect above observed treatment difference assuming observed standard deviations of two groups (i.e., 22.7 and 25.4) using a two-sided t-test with a 0.05 significance level.

# **Analysis Populations**

The intent-to-treat (ITT) population will include all randomized subjects who received IP.

The per protocol (PP) population is a subset of the ITT population, which will include all subjects who complete the study without major protocol deviations.

The safety population will include all subjects who received IP.

 Table 1
 Schedule of Visits and Examinations

| | Visit 1<br>Day -14 ± 2<br>Screening | Visit 2 Day 1 Baseline/ Randomization | Visit 3 Day 14 ± 2 Treatment | Visit 4<br>Day 28 ± 2<br>Treatment | Visit 5 Day 56 ± 4 Treatment/End of Assessments |
|---|---|---|---|---|---|
| Informed consent | X | | | | |
| Review inclusion/exclusion criteria | X | X | | | |
| Demographics | X | | | | |
| Medical and ocular history | X | | | | |
| Concomitant medication/review | X | X | X | X | X |
| Urine pregnancy test | X | | | | X |
| SANDE | X | X | X | X | X |
| VAS assessment of individual symptoms | | X | X | X | X |
| IP comfort assessment | | X | X | X | X |
| Best-corrected visual acuity | X | X | X | X | X |
| Biomicroscopy and external eye exam | X | X | X | X | X |
| Tear break-up time | X | X | X | X | X |
| Corneal fluorescein staining by zone | X | X | X | X | X |
| Anesthetized Schirmer's test | X | | | | |
| Dispense and provide instruction on administration/evaluate administration of run-in (vehicle) | X | | | | |
| Randomization | | X | | | |
| Dispense and provide instruction on administration investigational product (IP) | | X | | X | |
| Adverse event assessment | X | X | X | X | X |
| Run-in medication or IP return and accountability | | X | | X | X |

IP = investigational product; SANDE = Symptom Assessment in Dry Eye; VAS = visual analogue scale Subjects will receive their first dose of randomized IP in the clinic after successfully meeting inclusion criteria at Visit 2/Baseline.

# **TABLE OF CONTENTS**

| CLINIC | AL TRIAL PROTOCOL: SDP-4-CS202 | 1 |
|---------|---------------------------------------------------------------|----|
| SYNOPS | SIS | 2 |
| TABLE | OF CONTENTS | 9 |
| LIST OF | IN-TEXT TABLES | 13 |
| LIST OF | IN-TEXT FIGURES | 14 |
| LIST OF | ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 17 |
| 2. | STUDY OBJECTIVES | 19 |
| 2.1. | Primary Objective | 19 |
| 3. | INVESTIGATIONAL PLAN | 20 |
| 3.1. | Overall Study Design and Plan | 20 |
| 3.2. | Rationale for Study Design and Control Group | 20 |
| 3.3. | Study Duration and Dates | 21 |
| 4. | STUDY POPULATION SELECTION | 22 |
| 4.1. | Study Population | 22 |
| 4.2. | Inclusion Criteria | 22 |
| 4.3. | Exclusion Criteria | 22 |
| 5. | STUDY TREATMENT(S) | 26 |
| 5.1. | Description of Treatment(s) | 26 |
| 5.1.1. | Study Drug | 26 |
| 5.1.2. | Control | 26 |
| 5.2. | Selection, Timing and Administration of Dose for Each Patient | 26 |
| 5.3. | Method of Assigning Patients to Treatment Groups | 26 |
| 5.4. | Masking | 27 |
| 5.5. | Concomitant Therapy | 27 |
| 5.6. | Restrictions | 27 |
| 5.6.1. | Prohibited Medications and Treatments | 28 |
| 5.6.2. | Treatment Compliance | 29 |
| 5.7. | Packaging and Labeling. | 29 |
| 5.8. | Storage and Accountability | 29 |

| 5.9. | Investigational Product Dispensing and Retention at Study Site | 30 |
|---|---|---|
| 6. | STUDY PROCEDURES | 31 |
| 6.1. | Informed Consent | 31 |
| 6.2. | Demographics and Background Characteristics | 31 |
| 6.2.1. | Demographics | 31 |
| 6.2.2. | Medical/Ocular History | 31 |
| 6.2.3. | Medication History | 31 |
| 6.2.4. | Urine Pregnancy Test | 31 |
| 6.3. | Efficacy Assessments | 31 |
| 6.3.1. | Symptoms | 31 |
| 6.3.1.1. | SANDE (Symptom Assessment in Dry Eye) Questionnaire | 31 |
| 6.3.1.2. | Measurement of Individual Dry Eye Symptoms | 32 |
| 6.3.2. | Signs | 34 |
| 6.3.2.1. | Tear Break-up Time | 34 |
| 6.3.2.2. | Corneal Fluorescein Staining | 34 |
| 6.3.2.3. | Conjunctival Hyperemia | 35 |
| 6.4. | Adverse and Serious Adverse Events | 35 |
| 6.4.1. | Definition of Adverse Events | 35 |
| 6.4.1.1. | Adverse Event (AE) | 35 |
| 6.4.1.2. | Serious Adverse Event (SAE) | 35 |
| 6.5. | Relationship to Investigational Product | 36 |
| 6.6. | Recording Adverse Events | 36 |
| 6.7. | Reporting Adverse Events | 37 |
| 6.8. | Other Safety Assessments | 38 |
| 6.8.1. | Best-Corrected Visual Acuity | 38 |
| 6.8.2. | Biomicroscopy and External Eye Exam | 38 |
| 6.8.3. | Investigational Product Comfort Assessment | 39 |
| 6.9. | Screen Failures | 39 |
| 6.10. | Subject Withdrawal Criteria | 39 |
| 6.11. | Appropriateness of Measurements | 39 |
| 7. | STUDY ACTIVITIES | 40 |
| 7.1. | Visit 1 (Day -14 ± 2/Screening Visit) | 40 |

| 7.2. | Treatment Period (Day 1 to Day $56 \pm 4$ ) | 40 |
|---------|---------------------------------------------------------------|----|
| 7.2.1. | Visit 2 (Day 1/Confirmatory and Baseline/Randomization Visit) | 40 |
| 7.2.2. | Visit 3 (Day 14 ± 2) | 41 |
| 7.2.3. | Visit 4 (Day 28 ± 2) | 41 |
| 7.2.4. | Visit 5 (Day $56 \pm 4$ ) or Early Termination Procedures | 42 |
| 8. | QUALITY CONTROL AND ASSURANCE | 43 |
| 9. | STATISTICS | 44 |
| 9.1. | General Considerations | 44 |
| 9.2. | Determination of Sample Size | 44 |
| 9.3. | Analysis Populations | 44 |
| 9.3.1. | Intent-to-Treat (ITT) Population | 44 |
| 9.3.2. | Per Protocol (PP) Population | 44 |
| 9.3.3. | Safety Population | 45 |
| 9.4. | Demographics and Baseline Characteristics | 45 |
| 9.5. | Efficacy Endpoints and Analyses | 45 |
| 9.5.1. | Primary Efficacy Endpoint | 45 |
| 9.5.2. | Secondary Efficacy Endpoints | 45 |
| 9.5.3. | Efficacy Analyses | 45 |
| 9.6. | Safety Variables and Analysis | 46 |
| 9.6.1. | Safety Variables | 46 |
| 9.6.2. | Safety Analysis | 46 |
| 10. | ADMINISTRATIVE CONSIDERATIONS | 47 |
| 10.1. | Institutional Review Board (IRB) Approval | 47 |
| 10.2. | Ethical Conduct of the Study | 47 |
| 10.3. | Subject Information and Consent | 47 |
| 10.4. | Subject Confidentiality | 47 |
| 10.5. | Study Monitoring | 48 |
| 10.6. | Case Report Forms and Study Records | 49 |
| 10.7. | Protocol Deviations | 50 |
| 10.8. | Access to Source Documentation | 50 |
| 10.9. | Data Generation and Analysis | 50 |
| 10.9.1. | Retention of Data | 50 |

| 10.10. | Pub | lication and Disclosure Policy | 51 |
|---------|------|--------------------------------|----|
| 11. | REF | ERENCE LIST | 52 |
| APPENDI | X A. | SPONSOR SIGNATURES | 53 |
| APPENDI | ΧB | INVESTIGATOR'S SIGNATURE | 54 |

# LIST OF IN-TEXT TABLES

# LIST OF IN-TEXT FIGURES

| Figure 1: | Symptom Assessment in Dry Eye (SANDE) Questionnaire |
|---|---|
| Figure 2: | Division of the Corneal Surface for Measuring Fluorescein Uptake 33 |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE Adverse event

ANOVA Analysis of variance

BCVA Best-corrected visual acuity

BID Twice daily

CFR Code of Federal Regulations

CRA Clinical research associate

DED Dry eye disease

DSEK Descemet's stripping endothelial keratoplasty

eCRF Electronic case report form

eDC Electronic data capture

FDA Food and Drug Administration

GCP Good Clinical Practice

GLP Good Laboratory Practice

HCLE Human corneal limbal epithelial (cells)

HIPAA Health Information Portability and Accountability Act

IB Investigator's Brochure

ICH International Council for Harmonisation

IL Interleukin

IND Investigational New Drug

IOP Intraocular pressure

IP Investigational product

IRB Institutional Review Board

IV Intravenous

IWRS Interactive Web Response System

ITT Intent-to-treat

LASIK Laser-assisted in situ keratomileusis

LLOQ Lower limit of quantification

LRI Limbal relaxing incision

MedDRA Medical Dictionary for Regulatory Activities

MIGS Minimally invasive glaucoma surgery

MMP Matrix metalloprotease

MW Molecular weight

NF-κB Nuclear factor κB

NSAID Nonsteroidal anti-inflammatory drug

OHT Ocular hypertension

OU Both eyes

PP Per protocol

PRK Photorefractive keratectomy

SAE Serious adverse event

SANDE Symptom Assessment in Dry Eye

SDP-4 Silk-derived protein-4

SOP Standard operating procedure

SSNRI Selective serotonin norepinephrine reuptake inhibitors

SSRI Selective serotonin reuptake inhibitor

SUD Single-use dose

TEAE Treatment-emergent adverse event

TBUT Tear break-up time

TNF-α Tumor necrosis factor-alpha

US United States

VAS Visual Analog Scale

# 1. INTRODUCTION

Silk-derived protein-4 (SDP-4), also known as amlisimod, is a novel biotherapeutic being developed by SilkTech Biopharmaceuticals as a treatment for the signs and symptoms of dry eye disease (DED). Dry eye disease, as defined by the Tear Film and Ocular Surface Society (TFOS) Dry Eye Workshop (DEWS) II, is a "multifactorial disease of the ocular surface characterized by loss of homeostasis of the tear film and accompanied by ocular symptoms, in which tear film instability and hyperosmolarity, ocular surface inflammation and damage, and neurosensory abnormalities play etiological roles" (Craig et al., 2017).

The disease results in corneal irregularities that can create sight-limiting outcomes over time due to chronic inflammation governed, in part, by nuclear factor κB (NF-κB) signaling, which is thought to play a significant role in disease pathogenesis (Lan et al., 2012). Inflammatory mediators regulated by NF-κB, such as matrix metalloprotease (MMP)-9, tumor necrosis factor alpha (TNF-α), and interleukin (IL)-8 have been found in the tear fluid at high concentrations in patients exhibiting severe DED (Solomon et al., 2001; Smith et al., 2001). Furthermore, topical administration of MMP-9 to DED MMP-9-knockout mice subjected to DED inducing conditions via cholinergic blockade significantly increases corneal epithelial permeability, implicating MMP-9 in increased corneal epithelial disruption and damage (Pflugfelder et al., 2005). Collectively, these observations suggest a relationship between disruption of the corneal epithelium, increased secretion of MMP-9 through NF-κB signaling, and the signs and symptoms of DED.

Silk fibroin protein is the primary fibrous component of the *Bombyx mori* silkworm cocoon. *In vivo*, aqueous silk fibroin protein solution was successfully used to treat DED in a murine animal model, improving clinical outcomes (increased tear production, decreased corneal irregularity, inhibited epithelial cell detachment, and increased goblet cell density) and reducing inflammatory cytokine presence (intercellular adhesion molecule [ICAM]-1, vascular cell adhesion molecule [VCAM]-1, MMP-2 and MMP-9) (Kim et al, 2017).

Silk-derived protein (SDP) is a partially hydrolyzed population derived from the silk fiber protein fibroin with a molecular weight (MW) distribution of 2000-300,000 Daltons (Da). *In vitro* studies in immortalized hCLE cells subjected to scratch wound denudement demonstrated that aqueous SDP improved corneal epithelial wound healing through accelerated cell migration, proliferation and enhanced cell-matrix attachment (Abdel-Naby et al., 2017). Cultures treated with SDP displayed significant increases in cell-matrix focal adhesion formation and basement membrane adhesive strength compared to untreated cultures. *In vivo*, treatment with SDP accelerated the acute healing phase of injured rabbit corneal epithelial tissues, as shown by significantly increased epithelial migration rate, and produced a dose-dependent, 8-fold decrease in MMP-9.

Through a series of additional manufacturing steps, the subpopulation, SDP-4, is produced with a MW range of 10,000-30,000 Da. In nonclinical studies, SDP-4 has demonstrated a dual mechanism of action that both inhibits inflammation and physically improves the stability of the tear film. SDP-4 inhibits NF- $\kappa$ B driven expression of known dry eye inflammatory mediators produced by ocular surface cells, including MMP-9, TNF- $\alpha$ , and IL-8.

SilkTech has conducted nonclinical studies and one double-masked, randomized, vehicle-controlled, dose-response, parallel-group Phase II study to demonstrate the safety of SDP-4 in the treatment of DED. All 3 concentrations (0.1%, 1.0% and 3.0%) of SDP-4- were without major ocular or systemic safety issues in the Phase II study, with 1.0% concentration selected as the most appropriate for further clinical evaluation. A detailed description of the chemistry, pharmacology, and safety of SDP-4 is provided in the SDP-4 Investigator's Brochure.

# 2. STUDY OBJECTIVES

# 2.1. Primary Objective

The primary objective of this study is to assess the safety and efficacy of 1.0% SDP-4 Ophthalmic Solution in subjects with DED over an 8-week (56-day) treatment period.

# 3. INVESTIGATIONAL PLAN

# 3.1. Overall Study Design and Plan

This is a Phase 2, multicenter, double-masked, randomized, vehicle-controlled, dose-response, parallel-group study designed to evaluate the safety and efficacy of SDP-4 ophthalmic solution in subjects with moderate to severe DED in both eyes (OU) over an 8-week (56-day) treatment period.

Subjects will be randomized to 1.0% SDP-4 Ophthalmic Solution or vehicle in a 1:1 ratio in parallel groups. All investigational product (IP) (SDP-4 and vehicle) will be provided in single-use dose (SUD) containers packed in sealed foil pouches. Subjects, the Investigator, and all site personnel responsible for performing study assessments will remain masked to treatment assignment.

The IP will be administered via topical ocular instillation, one drop per eye, twice daily (BID) for 8 weeks (56 days). Both eyes will be treated with the same SUD at each dosing period. A 2-week screening/run-in period on BID vehicle will precede the 8-week randomized treatment period.

Subjects must have a Symptom Assessment in Dry Eye (SANDE) total score of  $\geq$  40 and  $\leq$  70 at Visit 1/Screening and Visit 2/Day 1 to enter the trial. For subjects with a qualifying SANDE score who meet all other inclusion/exclusion criteria, the eye with the lower tear break-up time (TBUT) at Visit 2/Day 1 will be designated as the study eye. In the event both eyes have the same TBUT scores, the eye with the lower Schirmer's test score at Visit 1 will be designated as the study eye. If both eyes have the same TBUT and Schirmer's test scores, the right eye will be designated as the study eye.

The study will consist of 5 clinic visits, 2 visits during the screening period and 3 on-treatment visits: Visit 1 (Day -14  $\pm$  2/Screening Visit), followed by the 2-week run-in period on BID vehicle, Visit 2 (Day 1/Confirmatory and Baseline/Randomization Visit), Visit 3 (Day 14  $\pm$  2), Visit 4 (Day 28  $\pm$  2), and Visit 5 (Day 56  $\pm$  4/End of Study Assessments).

See Table 1, Schedule of Visits and Examinations.

# 3.2. Rationale for Study Design and Control Group

It is hypothesized that by reducing pro-inflammatory mediators of DED, and providing a mucin replacement to enhance spreading and wetting of the tear film, SDP-4 will improve the symptoms of DED, as measured by the total SANDE score, and in the physical characteristics of the tear film measured by sign parameters, such as TBUT. The focus of this study is to demonstrate that enhanced patient selection will lead to a successful endpoint as measured by total SANDE score. Furthermore, the study will measure secondary endpoints including individual symptoms (itching, foreign body sensation, burning/stinging, fluctuating vision, eye dryness, eye discomfort, photophobia, and eye pain) and objective signs (TBUT, corneal fluorescein staining, and conjunctival hyperemia). 1.0% SDP-4 will be dosed topically BID versus vehicle to test the above stated hypothesis. The 1% SDP-4 concentration has been shown to produce maximal inhibition of NF-κB activity, and

combined with the physical properties of silk protein, is designed to provide for optimal clinical performance in the treatment of DED. The 8-week (56-day) treatment period provides for adequate assessment of the efficacy of the SDP-4 over time. The control being used in this study is the vehicle without the active ingredient of the drug product.

# 3.3. Study Duration and Dates

The duration of study treatment is 8 weeks (56 days). The overall duration of the study for each randomized subject is 10 weeks, which includes a 2-week screening/run-in period on vehicle and 8 weeks of treatment.

### 4. STUDY POPULATION SELECTION

# 4.1. Study Population

A total of 140 randomized subjects with DED (see Section 4.2) are planned, with 70 subjects assigned to 1.0% SDP-4 Ophthalmic Solution or vehicle.

### 4.2. Inclusion Criteria

Individuals must meet the following criteria at Screening (Visit 1/Day -14) and/or Visit 2/Day 1:

- 1. Willing and able to understand and sign an informed consent form prior to any study-related procedures.
- 2. Male or female patients 18 years of age or older.
- 3. Willing and able to follow study instructions, able to self-administer IP or have IP administered by a caregiver throughout the study period, and able to be present for the required study visits/assessments for the duration of the study.
- 4. Have DED in both eyes, as supported by a subject-reported history of daily symptoms of dry eye for  $\geq 6$  months prior to Visit 1/Screening requiring the use of artificial tears.
- 5. Total score  $\geq$  40 and  $\leq$  70 on the Symptom Assessment in Dry Eye (SANDE) questionnaire at Visits 1 and 2.
- 6. Tear break-up time (TBUT) of  $\leq$  6 seconds in both eyes at Visits 1 and 2.
- 7. Anesthetized Schirmer's test tear volume  $\geq 3$  mm and <10 mm in both eyes at Visit 1.
- 8. Best-corrected visual acuity (BCVA) of +0.7 logMAR or better in each eye as assessed by logMAR chart at Visits 1 and 2.
- 9. Female patients must be 1 year postmenopausal, surgically sterilized, or females of childbearing potential with a negative urine pregnancy test at Visit 1/Screening. Females of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include the use of at least one of the following: intrauterine device (IUD), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.

### 4.3. Exclusion Criteria

Individuals who meet any of the following criteria will be excluded from the study.

#### Ocular

- 1. Ocular surface corneal disease, other than DED.
- 2. Diagnosis of Sjögren's disease.
- 3. Lid margin disorder other than meibomian gland dysfunction (MGD) (e.g., active anterior blepharitis including staphylococcal, demodex or seborrheic; excessive lid

- laxity, floppy eyelid syndrome, ectropion, entropion) that in the Investigator's opinion could affect study parameters/assessments.
- 4. Presence of any ocular condition (e.g., pterygium) that in the Investigator's opinion could affect study parameters.
- 5. Any previous reconstructive or cosmetic eyelid surgery (e.g., blepharoplasty, ptosis repair, entropion/ectropion repair).
- 6. Any previous invasive glaucoma (e.g., trabeculectomy, shunt) and/or corneal surgery (e.g., penetrating keratoplasty, lamellar keratoplasty, Descemet's stripping endothelial keratoplasty [DSEK]).
- 7. Corneal refractive surgery (e.g., laser-assisted in situ keratomileusis [LASIK], photorefractive keratectomy [PRK], limbal relaxing incision [LRI]) within 12 months prior to Visit 1/Screening.
- 8. Cataract extraction, with or without minimally invasive glaucoma surgery (MIGS) or Yag capsulotomy, within 90 days prior to Visit 1/Screening.
- 9. Cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal within 30 days prior to Visit 1/Screening or planned during the study. If a subject has a punctal plug at Visit 1/Screening for ≥ 30 days and it falls out during the study, it should be replaced with a new plug of the same type.
- 10. Contact lens wear.

#### **Prior Medications**

- 11. Use of opioids within 90 days prior to Visit 1/Screening.
- 12. Use of isotretinoin (Accutane®) within 60 days prior to Visit 1/Screening.
- 13. Use of topical cyclosporine (Restasis<sup>®</sup>, Cequa<sup>®</sup>) or topical lifitegrast (Xiidra<sup>®</sup>) within 45 days prior to Visit 1/Screening.
- 14. Use of Visine® within 7 days prior to Visit 1/Screening.
- 15. Use of lid scrubs containing chemicals or baby shampoo within 14 days prior to Visit 1/Screening.
- 16. Use of any of the following medications within 30 days prior to Visit 1/Screening and throughout the study:
  - Topical ophthalmic corticosteroids or topical ophthalmic non-steroidal anti-inflammatory drugs (NSAIDs)
  - Autologous serum
  - Topical ophthalmic antibiotics or antivirals
  - Topical ophthalmic antihistamines or mast cell stabilizers
  - Topical ophthalmic medications for lowering of intraocular pressure (IOP) for treatment of glaucoma or ocular hypertension
  - Systemic immunosuppressive agents

- Systemic (i.e., oral, intravenous, intra-articular, intrathecal, epidural, or intramuscular) corticosteroids (dermatologic steroids other than around the eye or lid are allowed)
- Tetracycline compounds (tetracycline, doxycycline or minocycline) and systemic cyclosporine

### **Current Medications**

- 17. Any *changes* in the dosing of any chronically used systemic drug within 90 days prior to Visit 1/Screening and throughout the study period, including but not limited to the following (if a subject is taking any of the medications as needed (PRN), they must not be used within 7 days prior to Visit 1/Screening and discontinued throughout the study period):
  - Anticholinergics
  - Antidepressants including selective serotonin reuptake inhibitors (SSRIs), selective serotonin norepinephrine reuptake inhibitors (SSNRIs), tricyclics, and benzodiazepines
  - Antihistamines
  - Systemic H1-receptor antagonists
  - β-adrenoceptor antagonists
  - Calcium channel blockers
- 18. Any *changes* in the dosing of aspirin and aspirin-containing products within 30 days prior to Visit 1/Screening and throughout the study period.

#### General

- 19. Stevens-Johnson syndrome.
- 20. History of immunodeficiency disorder, HIV, positive hepatitis B, C, or evidence of acute active hepatitis A (anti–HAV IgM).
- 21. History of organ or bone marrow transplant.
- 22. History of graft versus host disease (GvHD).
- 23. Systemic lupus erythematosus.
- 24. Chronic pain syndrome (e.g., fibromyalgia).
- 25. Systemic signs of infection (e.g., fever or current treatment with antibiotics).
- 26. Serious systemic disease or uncontrolled medical condition that in the judgment of the Investigator could confound study assessments or limit compliance, including, but not limited to, severe cardiopulmonary disease, poorly controlled hypertension, and/or poorly controlled diabetes.
- 27. Known history of alcohol and/or drug abuse within 12 months prior to Visit 1/Screening that, in the opinion of the Investigator, may interfere with study

- compliance, outcome measures, safety parameters, and/or the general medical condition of the subject.
- 28. Known allergy or contraindication to any component of IP formulation or diagnostic agents.
- 29. Participation in any drug or device clinical investigation within 30 days prior to Visit 1/Screening and/or during the period of study participation.
- 30. Screening and enrollment of more than one individual who resides in the same household.
- 31. Screening and enrollment of employees of the clinical site.
- 32. Screening and enrollment of subjects who participated in the SDP-4-CS201 trial.

# 5. STUDY TREATMENT(S)

# **5.1.** Description of Treatment(s)

# 5.1.1. Study Drug

SDP-4 Ophthalmic Solution is a non-preserved aqueous solution of SDP-4 for topical ophthalmic use and will contain the active substance (SDP-4) and polysorbate-80, sodium acetate trihydrate, glacial acetic acid, magnesium chloride hexahydrate, and dextrose monohydrate.

#### **5.1.2.** Control

The vehicle solution will be the same as the SDP-4 except for the omission of the active substance (SDP-4).

All subjects who meet study entry criteria at Screening/Visit 1 (Day -14  $\pm$  2) will receive a supply of vehicle solution prior to randomization to the double-masked study to be administered during the 14-day ( $\pm$  2) screening/run-in period.

# 5.2. Selection, Timing and Administration of Dose for Each Patient

Subjects will be randomized to treatment with 1.0% SDP-4 Ophthalmic Solution or vehicle which will be administered to each eye BID, approximately 12 hours apart, for 56 days.

Subjects (or their caregiver, if the subject is not able to self-administer the IP) will administer IP topically OU BID for 56 days. At the Screening and Baseline visits, site personnel will instruct the subject (or caregiver) in topical ocular drop administration procedures. After instilling a drop in each eye, the used single-unit dose (SUD) vials should be stored in the storage container provided by site personnel and placed back in the box.

Twice each day, approximately 12 hours apart, the subject (or caregiver) will open a new SUD and administer 1 drop to each eye from the same vial, store the used SUD vial in the foil pouch, and place it in the box (or storage container) for return to the clinical site so accountability can be documented in the source document and electronic case report form (eCRF). All IP, including the box, used SUDs/foil pouches and any unopened SUD vials will be returned to the clinical site where the used and unopened IP will be documented at Visits 2, 4 and 5.

# 5.3. Method of Assigning Patients to Treatment Groups

Subjects will be randomized in a 1:1 ratio to 1.0% SDP-4 or vehicle in parallel groups. A computer-generated randomization code for allocating the solutions will be prepared by an independent unmasked biostatistician not involved in the day-to-day running of the study.

If subjects meet eligibility criteria at Screening (Visit 1/Day -14) and Visit 2/Day 1 (see Section 4 for eligibility criteria), subjects will be randomly assigned to IP at Visit 2. Clinical sites will utilize the Interactive Web Response System (IWRS) to assign kits to subjects. The IP kit randomization number will be recorded in the subject's eCRF.

# 5.4. Masking

The study will be double-masked. SDP-4 and vehicle will be provided in SUD vials packed in sealed foil pouches which are enclosed in a box and dispensed in one-month supplies at Visits 2 and 4. Subjects, the Investigator, and all site personnel responsible for performing study assessments will remain masked to treatment assignment.

Should it be necessary to unmask a subject's treatment assignment in case of emergency, the Investigator may obtain the treatment code for a given randomized subject from the IWRS. The treatment code is to be obtained only if a medical emergency exists and knowledge of the medication being taken will influence the medical management of the subject.

The following procedure should be followed:

- 1. The Investigator should contact the Medical Monitor via phone immediately before unmasking a subject, unless it is not possible to do so without risk to the subject.
- 2. The Investigator should document the serious adverse event (SAE), if applicable, and justification for unmasking in the eCRF.
- 3. The subject may continue to participate in the study to be followed for safety at the Investigator's discretion. If the subject is to be discontinued from study participation, then ALL procedures described in the Early Discontinuation Visit (Section ) should be completed.
- 4. The Investigator should contact the Medical Monitor at Safety@silk-tech.com within 24 hours with the randomization number, details of the adverse event (AE) or SAE, any action taken, and whether the subject is continuing in the study.

# 5.5. Concomitant Therapy

Therapy considered necessary for the subject's welfare that will not interfere with the evaluation of the IP may be given at the discretion of the Investigator and in consultation with the Medical Monitor. If there is any question as to whether the medication may interfere, the Investigator should contact the Sponsor.

Permitted steroid medications include intranasal, inhaled, dermatologic (other than those around the eye or lid), or peri-anal steroids.

Whenever possible, medications should be administered in dosages that remain stable throughout the study duration. All concomitant medications will be recorded in the eCRF.

### 5.6. Restrictions

The Medical Monitor should be notified before prohibited medication or therapy is administered, unless the safety of the subject requires immediate action. The decision to administer a prohibited medication or therapy should be done with the safety of the subject as the primary consideration. The Medical Monitor should be contacted to determine the permissibility of a specific medication or therapy and whether or not the subject should continue with study participation.

# 5.6.1. Prohibited Medications and Treatments

In addition to the exclusion listed in Section 4.3, the following medications are prohibited as specified:

Within 60 days prior to Visit 1/Screening and throughout the study duration:

• Use of isotretinoin (Accutane)

Within 45 days prior to Visit 1/Screening and throughout the study duration:

• Use of topical cyclosporine (Restasis, Cequa) or topical lifitegrast (Xiidra)

Within 30 days prior to Visit 1/Screening and throughout the study duration:

- Topical ophthalmic corticosteroids or topical ophthalmic NSAIDs
- Autologous serum
- Topical ophthalmic antibiotics or antivirals
- Topical ophthalmic antihistamines or mast cell stabilizers
- Topical ophthalmic medications for lowering of IOP for treatment of glaucoma or OHT
- Systemic immunosuppressive agents other than corticosteroids
- Systemic (oral, intravenous, intra-articular, intrathecal, epidural or intramuscular) corticosteroids
- Tetracycline compounds (e.g., tetracycline, doxycycline or minocycline) and systemic cyclosporine

Any *change* in the dosing of the following within 90 days prior to Visit 1/Screening and throughout the study duration:

- Anticholinergics
- Antidepressants including selective serotonin reuptake inhibitors (SSRIs), selective serotonin norepinephrine reuptake inhibitors (SSNRIs), tricyclics, and benzodiazepines
- Antihistamines
- Systemic H1-receptor antagonists
- β-adrenoceptor antagonists
- Calcium channel blockers

Any *change* in the dosing of the following within 30 days prior to Visit 1/Screening and throughout the study duration:

• Aspirin and aspirin-containing products

The following procedures are prohibited as specified:

Any previous:

- Reconstructive or cosmetic eyelid surgery (e.g., blepharoplasty, ptosis repair, entropion/ectropion repair)
- Invasive glaucoma (e.g., trabeculectomy, shunt) and/or corneal surgery (e.g., penetrating keratoplasty, lamellar keratoplasty, DSEK)

Within 12 months prior to Visit 1/Screening:

• Corneal refractive surgery (e.g., LASIK, PRK, LRI)

Within 90 days prior to Visit 1/Screening:

• Cataract extraction, with or without MIGS or Yag capsulotomy

Within 30 days prior to Visit 1/Screening and throughout the study period:

• Cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal. If a subject has a punctal plug at Visit 1/Screening for ≥ 30 days and it falls out during the study, it should be replaced with a new plug of the same type.

Contact lens wear prior to and during the study is prohibited.

## **5.6.2.** Treatment Compliance

Treatment compliance will be monitored by IP accountability throughout the study. The amount of used and unused run-in vehicle returned at Visit 2/Day 1 and used and unused randomized IP returned at Visit 4/Day 28 and Visit 5/Day 56 will be documented by site personnel.

# 5.7. Packaging and Labeling

The IP will be filled into BFS containers composed of low-density polyethylene (LDPE). The individual cartridges of 5 SUD vials will be seal packed into a foil pouch. The foil-wrapped cartridges will be packaged 7 at a time into a cardstock storage box that will contain a total of 35 SUD vials for the 2-week run-in period. The foil-wrapped pouches will be packaged 12 at a time into a cardstock storage box that will contain a total of 60 SUD vials dispensed at Visit 2 and 13 at a time into a cardstock storage box that will contain a total of 65 SUD vials dispensed at Visit 4 during the randomized treatment period. A label bearing the required IP labeling information per Code of Federal Regulations (CFR) Part 312, Section 312.6 will be added on the outside of the foil wrapping and the outside of the IP storage box.

# 5.8. Storage and Accountability

The IP should be stored at a controlled temperature at 15°- 25°C (59°-77°F) in a secured area. A temperature log will be maintained at each clinical site. Subjects should be instructed to store IP at home at room temperature. After opening a foil pouch, the remaining SUDs should be stored in the pouch until used. Subjects will retain all used and unused IP materials (SUD vials, foil pouches, boxes) to return to the site.

# 5.9. Investigational Product Dispensing and Retention at Study Site

At Visit 1/Screening, if the eligibility criteria are met, vehicle solution for the screening/run-in period will be dispensed to the subject with instructions to return the used and unused IP at Visit 2/Day 1. When the run-in study materials are returned by the subject, accountability will be performed and the box will be retained at the site in a secured location.

At Visit 2/Day 1, Kit 1 will be dispensed after the subject is randomized. Kit 2 will remain in a secured location at the site. The subject will be instructed to return the box along with all used and unused IP study materials at Visit 4/Day 28.

At Visit 4/Day 28, when Kit 1 is returned by the subject, accountability will be performed, and the kit will be retained at the site in a secured location. The site will dispense Kit 2 to the subject according to randomization number with instructions to return the box along with used and unused IP study materials at Visit 5/Day 56.

At Visit 5/Day 56, when Kit 2 is returned by the subject, accountability will be performed, and the kit will be retained at the site in a secured location for the clinical research associate (CRA) to perform IP accountability and reconciliation. At the end of the study, the site or CRA will ship the IP study materials back to the packager for destruction.

### 6. STUDY PROCEDURES

# 6.1. Informed Consent

Prior to entry into the study or initiation of any study-related procedures, the subject must read, sign, and date the current Institutional Review Board (IRB)-approved version of the informed consent form. A full discussion of informed consent is presented in Section 10.3.

# 6.2. Demographics and Background Characteristics

### 6.2.1. Demographics

Demographic information including age, gender, race, ethnicity, and date of informed consent will be recorded.

# 6.2.2. Medical/Ocular History

Clinically significant medical and ocular history will be documented and will include any previously diagnosed ocular abnormalities and ocular surgeries, including laser and non-laser procedures.

# **6.2.3.** Medication History

All current medications (prescription and over-the-counter) taken at Screening, 90 days prior to Screening, and throughout the course of the study will be recorded in the Concomitant Medications page of the eCRF. Information regarding the dates of first and last dose, site of dosing (e.g., right eye, left eye, OU, systemic), and the reason the medication is being taken must be recorded in the eCRF.

#### **6.2.4.** Urine Pregnancy Test

A urine pregnancy test will be performed at Visit 1/Screening and repeated at Visit 5/Day 56 or the Early Discontinuation Visit for women of childbearing potential only.

# **6.3.** Efficacy Assessments

Efficacy will be measured by assessment of DED symptoms (SANDE total score, individual symptoms rated on a visual analogue scale [VAS]: itching, foreign body sensation, burning/stinging, fluctuating vision, eye dryness, eye discomfort, photophobia, and eye pain), and signs (TBUT, corneal fluorescein staining, and conjunctival hyperemia). All efficacy assessments will be conducted at the timepoints shown on the Schedule of Visits and Examinations (Table 1).

# **6.3.1.** Symptoms

#### 6.3.1.1. SANDE (Symptom Assessment in Dry Eye) Questionnaire

The SANDE contains two questions regarding the frequency and severity of DED symptoms as shown in Figure 1.

# Figure 1: Symptom Assessment in Dry Eye (SANDE) Questionnaire

### 1. Frequency of symptoms:

Please place a mark on the line to indicate how often, on average, your eyes feel dry and/or irritated:



# 2. Severity of symptoms:

Please place a mark on the line to indicate how severe, on average, you feel your symptoms of dryness and/or irritation are:



Source: Schaumberg et al., 2007

The frequency and severity scores (SANDE) will be recorded in the eCRF. The total score is the square root of the frequency score times the square root of the severity score (range 0-100) and will be calculated by the electronic data capture (eDC) system.

## **6.3.1.2.** Measurement of Individual Dry Eye Symptoms

The following individual symptoms of DED will be evaluated using a separate VAS scale for each symptom and will include: itching, foreign body sensation, burning/stinging, fluctuating vision, eye dryness, eye discomfort, photophobia, and eye pain.

The subject will be asked to make a mark on the line to indicate how he/she feels about each symptom since the last visit.

### Itching



Doesn't itch at all

Want to scratch my eyes out





Don't feel like I have something in my eye

Feels like I have sand in my eye

# **Burning/Stinging**



Doesn't burn/sting at all

Severe

# **Fluctuating Vision**



Vision is fine

Vision constantly changes

# **Eye Dryness**



Not dry at all Extremely dry

## **Eye Discomfort**



Very comfortable

Extremely uncomfortable

### **Photophobia**



Not sensitive to light

Extremely sensitive to light

# Eye Pain



No eye pain Need pain medicine

The score for each symptom will be recorded in the eCRF.

### **6.3.2.** Signs

### 6.3.2.1. Tear Break-up Time

The tear film will be observed under the slit-lamp and timed until the tear film breaks up (i.e., tiny dry spots develop) (Nichols et al., 2004). The procedure is conducted 2 times for each eye and the TBUT for each is measured in seconds and recorded in the eCRF. The average for each eye will be calculated by the eDC system. Consult the Study Reference Manual for specific details regarding the evaluation procedures.

# 6.3.2.2. Corneal Fluorescein Staining

Following evaluation of TBUT, corneal fluorescein staining using a Wratten #12 filter (or equivalent) will be measured using the National Eye Institute (NEI) standardized grading system to grade each of the 5 areas of the cornea on a 0-3 scale as shown in Figure 2 (range:

0-15) (Lemp, 1995). Consult the Study Reference Manual for specific details regarding the evaluation procedures.

Figure 2: Division of the Corneal Surface for Measuring Fluorescein Uptake



Source: Lemp, 1995

## 6.3.2.3. Conjunctival Hyperemia

Conjunctival hyperemia will be graded during the slit-lamp examination using the McMonnies photographic scale (McMonnies and Chapman, 1987a; McMonnies and Chapman, 1987b). This photographic reference scale consists of 6 levels or grades of conjunctival hyperemia (0 = none, 5 = severe). Please note that these were designed for contact lens wearers, but validated for non-contact lens wearers (McMonnies and Ho, 1991). Consult the Study Reference Manual for specific details regarding the evaluation procedures.

## **6.4.** Adverse and Serious Adverse Events

#### **6.4.1.** Definition of Adverse Events

### 6.4.1.1. Adverse Event (AE)

An AE is any untoward medical occurrence in a clinical study subject administered an IP that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IP, whether or not considered related to this IP.

Note: IP in this study refers to 1.0% SDP-4 and to the vehicle (control).

Medical conditions/diseases present before starting the investigational treatment are only considered AEs if they worsen after starting the investigational treatment. Abnormal test results constitute AEs only if they induce clinical signs or symptoms, are considered clinically significant, or require therapy.

The occurrence of AEs should be sought by open-ended questioning of the subject at each visit during the study. At each clinic visit, study personnel should ask the following question: "Have you had any problems since your last visit?" Adverse events also may be detected when they are volunteered by the subject during or between visits or through study assessments.

#### **6.4.1.2.** Serious Adverse Event (SAE)

An SAE is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening or sight-threatening

Note: The term "life-threatening" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.

- Results in persistent or significant disability/incapacity (excluding progression/outcome of the disease under study)
- Is a congenital anomaly/birth defect
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Is medically significant; i.e., defined as an event that jeopardizes the health of the subject or may require medical or surgical intervention to prevent one of the outcomes listed above

Treatment on an outpatient emergency basis that does not result in hospital admission, or a hospitalization that is elective or is a preplanned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since the start of the study, is not considered an SAE.

All SAEs that are ongoing at the time of completion or discontinuation from the study will be followed until stabilization or resolution of the event.

# 6.5. Relationship to Investigational Product

The relationship of AEs to the IP should be assessed by the Investigator using the definitions below.

**Not suspected:** The temporal relationship of the event to the IP makes a causal relationship unlikely, or, other drugs, therapeutic interventions or underlying conditions provide a sufficient explanation for the observed event.

**Suspected:** The temporal relationship of the event to the IP makes a causal relationship possible or other drugs, therapeutic interventions or underlying conditions do not provide a sufficient explanation for the observed event.

If there is any valid reason, even if undetermined, for suspecting a possible cause-and-effect relationship between the IP and the occurrence of the AE, then the AE should be considered "suspected."

If the relationship between the AE/SAE and the IP is determined by the Sponsor to be "suspected" the event will be considered to be related to the IP for the purposes of expedited regulatory reporting.

# **6.6.** Recording Adverse Events

Adverse events spontaneously reported by the subject and/or in response to an open question from the study personnel or revealed by observation, regardless of severity or potential association with the IP or study procedures, will be recorded in the eCRF. Changes from
baseline assessments that are part of the disease being studied will not necessarily be recorded as AEs unless the Investigator deems them as such. Investigators are advised to consider reporting a visual acuity decrease of 3 lines EDTRS (15 letters) or greater as an AE. If ongoing at the time of the subject's last study visit, Investigators should follow the event until the subject has returned to baseline or the event has resolved.

All AEs that occur following consent and until the final study visit (Visit 5/Day 56) should be collected and recorded on the AE eCRF page. AEs that occur during the screening/run-in period (Visit  $1/\text{Day}-14 \pm 2$  to Visit 2/Day 1) will be summarized separately from AEs that occur from the first dose of double-masked treatment on Day 1 to the Day 56 Visit or Early Discontinuation. Serious adverse events (SAEs) will be followed until the event is resolved or stabilized.

The AE term should be reported in standard medical terminology when possible. For each AE, the Investigator will evaluate and report the following:

- Onset (date)
- Resolution (date)
- Severity grade (mild, moderate, severe)
- Relationship to IP (not suspected, suspected)
- Action taken (none, IP temporarily interrupted, IP permanently discontinued; concomitant medication taken; hospitalization/prolonged hospitalization; other)
- Serious outcome (yes/no)

The severity grade should be determined by the Investigator using the definitions below:

- Mild: Discomfort noticed but no disruption of normal daily activity
- Moderate: Discomfort sufficient to cause interference with normal daily activity
- Severe: Incapacitating, with inability to perform normal activities

It is important to distinguish between serious and severe AEs. Severity is a measure of intensity (as defined directly above) whereas seriousness is defined by the criteria under Section 6.4.1.2. An AE of severe intensity may not be considered serious.

Should a pregnancy occur, it must be reported and recorded on the pregnancy form. Pregnancy in itself is not regarded as an AE unless there is a suspicion that an IP may have interfered with the effectiveness of a contraceptive medication. The subject will stop using the IP, be withdrawn from the study, and followed through conclusion of pregnancy. The outcome of all pregnancies (spontaneous miscarriage, elective termination, normal birth or congenital abnormality) must be followed up and documented.

# 6.7. Reporting Adverse Events

All AEs (suspected and not suspected) will be recorded following consent and until the final study visit, Visit 5/Day 56. Any SAEs "suspected" to be related to the IP and discovered by the Investigator at any time after the study should be reported.

Any SAE that occurs must be reported within 24 hours of its occurrence or within 24 hours of learning of its occurrence by entering the information in the appropriate eCRF page in the EDC system. Recurrent episodes, complications, or progression of the initial SAE must be reported as follow-up to the original episode within 24 hours of the Investigator receiving the information. Information about all SAEs will be collected and recorded on the SAE form. All pertinent medical records and information collected during the treatment and follow-up of the subject should be maintained at the site with a copy emailed to <a href="Safety@silk-tech.com">Safety@silk-tech.com</a> only if requested and after thorough de-identification/removal of all personal health information (PHI). The Investigator must assess the SAE relationship to the IP/study treatment and severity and complete the SAE form. Silk Technologies may request additional information. Follow-up information (e.g., discharge summary) will be retained in the subject's chart and a copy will be emailed to Safety@silk-tech.com.

In addition, all SAEs should be recorded on the Adverse Event eCRF page with the serious question marked "Yes".

All subjects who experience an SAE should be followed clinically and undergo the appropriate diagnostic evaluations until stabilization or resolution of the event.

It is the Investigator's responsibility to notify the approving IRB of any site-specific SAEs per the IRB's reporting requirements.

Silk Technologies will report all SAEs to the United States (US) Food and Drug Administration (FDA) on the appropriate schedule depending if the event is IP related or not IP related, expected or unexpected (based on the available information in the IB).

Any death occurring during the study and follow up period should be reported as an SAE. For any death occurring through the end of the study, regardless of the degree of relationship to IP, the SAE resulting in the death must be reported to Silk Technologies or designee. A death occurring after completion of the study does not require completion of the SAE form.

# **6.8.** Other Safety Assessments

#### **6.8.1.** Best-Corrected Visual Acuity

Best-corrected visual acuity (BCVA) measurement will be performed in each eye at all study visits with the logMAR eye chart using the subject's best corrective lens prescription eyeglasses or trial frame lenses, if applicable. The subject's BCVA must be determined (via refraction) if corrected or uncorrected visual acuity is not logMAR 0.0 (equivalent to 20/20). This refraction must be used for all VA assessments for the duration of the study. The subject must wear the same glasses/trial frame, if applicable, at each visit. Ambient room lighting should be consistent for a given subject throughout the study period. Consult the Study Reference Manual for specific details regarding the evaluation procedures.

## **6.8.2.** Biomicroscopy and External Eye Exam

A slit-lamp examination will be conducted at each study visit to assess the anterior ocular structures, including lid, cornea, conjunctiva, anterior chamber, iris, lens, and posterior capsule (if pseudophakic). Abnormalities will be documented. Consult the Study Reference Manual for specific details regarding the evaluation procedures.

## 6.8.3. Investigational Product Comfort Assessment

Subjects will rate the comfort of IP instillation according to the following 4-point scale:

- 0 = No discomfort
- 1 = Mild discomfort
- 2 = Moderate discomfort
- 3 =Severe discomfort

#### 6.9. Screen Failures

A screen failure is a subject who has given informed consent but failed to meet the inclusion criteria or met at least 1 of the exclusion criteria, and has not been randomized into the study. Based on Investigator discretion and Sponsor approval, subjects who initially failed to meet the inclusion/exclusion criteria may be rescreened at a later time if their eligibility status has changed. The subject will retain the same subject identification number that he/she was assigned at the first screening.

## 6.10. Subject Withdrawal Criteria

The following are the criteria for considering withdrawal from the study:

- Withdrawal of subject consent. The subject may request for any reason at any time to be withdrawn from the study.
- Investigator/Sponsor decision (prohibited medication, compliance, etc.)
- The Sponsor terminates the study.

If a subject withdraws from the study, the reason for withdrawal will be recorded in the eCRF.

If a study subject fails to attend a study visit at any point during the study period, every effort should be made to keep the subject in the study and conduct all study visits as scheduled; all attempts to contact the subject must be documented. If the subject relocates during the study period, the CRO should be contacted to determine if there is a possibility that the subject could continue at another clinical site.

# 6.11. Appropriateness of Measurements

The efficacy and safety assessments in this study are standard for ophthalmologic investigations, and their reliability, accuracy, and relevance is well established. Collection of AEs to monitor drug safety is standard in clinical studies.

#### 7. STUDY ACTIVITIES

Table 1 provides a tabular summary of all scheduled visits and procedures to be performed during the clinical study.

## 7.1. Visit 1 (Day -14 $\pm$ 2/Screening Visit)

Procedures performed at Screening, Visit  $1/\text{Day} - 14 \pm 2$  will include the following:

- Obtain written informed consent
- Inclusion/exclusion criteria
- Demographics
- Medical and ocular history
- Concomitant medication review
- Urine pregnancy test (women of childbearing potential only)
- SANDE
- BCVA (logMAR)
- Biomicroscopy/external eye exam
- TBUT
- Corneal fluorescein staining
- Anesthetized Schirmer's test
- Re-review inclusion/exclusion criteria
- Dispense run-in medication/provide instruction on administration/in-clinic administration/evaluate administration
- AE assessment

Eligible subjects must have daily symptoms of DED for  $\geq 6$  months, a total score  $\geq 40$  and  $\leq 70$  on the SANDE questionnaire, history of artificial tear use in the 30 days prior to Screening, TBUT  $\leq 6$  seconds in both eyes, and anesthetized Schirmer's test tear volume  $\geq 3$  mm and  $\leq 10$  mm in both eyes.

# 7.2. Treatment Period (Day 1 to Day $56 \pm 4$ )

## 7.2.1. Visit 2 (Day 1/Confirmatory and Baseline/Randomization Visit)

Procedures performed at Visit 2/Day 1 include:

- Concomitant medication review
- SANDE
- Individual symptom assessment (VAS)
- IP comfort assessment

- BCVA (logMAR)
- Biomicroscopy/external eye exam
- TBUT
- Corneal fluorescein staining
- Review inclusion/exclusion criteria
- Randomize eligible subjects
- Dispense IP/provide instruction on administration
- Self-administration of first dose of randomized IP in the clinic
- AE assessment
- Run-in medication accountability

## 7.2.2. Visit 3 (Day $14 \pm 2$ )

Procedures performed at Visit 3/Day  $14 \pm 2$  include:

- Concomitant medication review
- SANDE
- Individual symptom assessment (VAS)
- IP comfort assessment
- BCVA (logMAR)
- Biomicroscopy/external eye exam
- TBUT
- Corneal fluorescein staining
- AE assessment

### 7.2.3. Visit 4 (Day $28 \pm 2$ )

Procedures performed at Visit 4/Day  $28 \pm 2$  include:

- Concomitant medication review
- SANDE
- Individual symptom assessment (VAS)
- IP comfort assessment
- BCVA (logMAR)
- Biomicroscopy/external eye exam
- TBUT
- Corneal fluorescein staining

- Dispense IP/provide instruction on administration
- IP accountability
- AE assessment

## 7.2.4. Visit 5 (Day $56 \pm 4$ ) or Early Termination Procedures

Procedures performed at Visit 5/Day  $56 \pm 4$  include:

- Concomitant medication review
- SANDE
- Individual symptom assessment (VAS)
- IP comfort assessment
- BCVA (logMAR)
- Biomicroscopy/external eye exam
- TBUT
- Corneal fluorescein staining
- Urine pregnancy test (women of childbearing potential only)
- AE assessment
- IP accountability

## 8. QUALITY CONTROL AND ASSURANCE

Silk Technologies and/or their contracted agents utilize standard operating procedures (SOPs) designed to ensure that research procedures and documentation are consistently conducted/prepared to the highest quality standards. These SOPs require compliance with FDA regulations and the International Council for Harmonisation (ICH) Good Clinical Practice (GCP) guidance.

The study will be monitored by CRAs/monitors to verify that the rights and well-being of human subjects are being protected, the reported data are accurate, complete, and verifiable, and that the conduct of the study is in compliance with the currently approved protocol, with ICH GCP, and with the applicable regulatory requirements.

To ensure compliance with GCP and all applicable regulatory requirements, Silk Technologies or its agents may conduct a quality assurance audit at any time during or after completion of a study. The Investigator will be given adequate notice if s/he is selected for an audit. The audit will include, but is not limited to: a review of all informed consent forms, medical records, and regulatory documentation; an assessment of study conduct and protocol compliance; and a review of the study materials receipt, storage, and administration. At the conclusion of an audit, the auditor will conduct a brief meeting with the Investigator to review the findings of the audit.

#### 9. STATISTICS

## 9.1. General Considerations

This is a Phase 2, multicenter, randomized, double-masked, vehicle-controlled, parallel group study to evaluate the safety and efficacy of 1.0% SDP-4 ophthalmic solution in subjects with DED.

Subjects with DED are planned to be randomized to SDP-4 (1.0%) or vehicle in a 1:1 ratio, with 70 subjects randomized to each group.

A biostatistician will perform statistical analyses as agreed with the Sponsor according to the Statistical Analysis Plan (SAP).

All continuous study assessments will be summarized by treatment and visit (as applicable) using descriptive statistics (n, mean, median, standard deviation, minimum, and maximum). All categorical study assessments will be summarized by treatment and visit (as applicable) using frequency counts and percentages.

All study data will be listed by treatment, subject, and visit (as applicable).

The unit of analysis for efficacy will be the study eye.

Efficacy analysis will be conducted on the intent-to-treat (ITT) population (primary efficacy analysis) and the per protocol (PP) population (secondary efficacy analysis). Safety analyses will be performed using the safety analysis population. Definitions for the analysis populations may be found in Section 9.3.

# 9.2. Determination of Sample Size

Based on results from SDP-4-CS201, a treatment difference of 12.2 units SANDE total score mean change from baseline at Day 56 was observed in the subgroup population meeting the Total SANDE score  $\geq$  40 and  $\leq$  70. A sample size of 70 subjects per treatment group will have 84.5% power to detect above observed treatment difference assuming observed standard deviations of the two groups (i.e., 22.7 and 25.4) using a two-sided t-test with a 0.05 significance level.

# 9.3. Analysis Populations

#### 9.3.1. Intent-to-Treat (ITT) Population

The ITT population will include all randomized subjects who received IP. This population will be the primary population for efficacy analyses and will be used to summarize all efficacy variables and will summarize subjects as randomized.

#### 9.3.2. Per Protocol (PP) Population

The PP population is a subset of the ITT population, which will include all subjects who complete the study without major protocol deviations. This population will be the secondary population for efficacy analyses and will be used to summarize a subset of efficacy variables. The PP population will summarize subjects as treated.

#### 9.3.3. Safety Population

The safety population will include all subjects who received IP. This population will be used to summarize safety variables and will summarize subjects as treated.

## 9.4. Demographics and Baseline Characteristics

Subject demographic and baseline characteristics will be summarized in tables. Summary tables will be supported with individual subject data listings.

## 9.5. Efficacy Endpoints and Analyses

## 9.5.1. Primary Efficacy Endpoint

Mean change from baseline in total SANDE score at Visit 5/Day 56

### 9.5.2. Secondary Efficacy Endpoints

- Mean and mean change from baseline at each visit for each of the following evaluations:
  - Corneal fluorescein staining (combined and each zone)
  - TBUT
  - Conjunctival hyperemia
  - Individual symptom VAS scores, separately for each symptom

#### SANDE

- Mean change from baseline in total SANDE score at each visit
- Mean total SANDE score at each visit
- Mean and mean change from baseline in each component of SANDE at each visit

#### 9.5.3. Efficacy Analyses

The primary efficacy endpoint (SANDE) will be summarized using continuous summary statistics by treatment group and visit. The primary analysis will utilize a repeated measures mixed model where the dependent variable is the change from baseline score, treatment group is a fixed effect, baseline score is a covariate, and visit is a repeated measure on subject. The repeated measures mixed model is utilized to account for the effect of missing data under the assumption that the data are missing at random. Least squares means will be used to test SDP-4 to vehicle. Sensitivity analyses for the primary endpoint will be performed using last observation carried forward (LOCF) as well as observed data only.

The planned analyses for all efficacy outcomes will be described in detail in the SAP, which will be finalized prior to database lock.

## 9.6. Safety Variables and Analysis

#### 9.6.1. Safety Variables

Safety variables are as follows:

- Ocular and non-ocular AE monitoring
- BCVA
- Biomicroscopy
- IP comfort assessment

## 9.6.2. Safety Analysis

Safety and IP comfort data will be presented in tables of descriptive statistics and frequency distribution. All summary tables will be supported with individual subject data listings.

AEs that occur during the screening/run-in period (Visit  $1/\text{Day-}14 \pm 2$  to Visit 2/Day 1) will be summarized separately from AEs that occur from the first dose of double-masked treatment on Day 1 to the Day 56 Visit or Early Discontinuation.

The primary safety analysis will summarize ocular and non-ocular treatment-emergent adverse events (TEAEs) using discrete summaries at the subject level by system organ class and preferred term for each treatment group. A TEAE will be defined as occurring after the first dose of IP. Serious adverse events (SAEs) and treatment-related ocular and non-ocular TEAEs will be summarized similarly. Ocular and non-ocular TEAEs will also be summarized by severity.

Biomicroscopy and dilated indirect ophthalmoscopy measures will be summarized by tabulating the distribution of score shifts between baseline and post-baseline assessments

Best-corrected visual acuity (BCVA; logMAR) will be summarized at each visit, using continuous and discrete summary statistics, including change from baseline and the proportion of study eyes with pre-defined increases from baseline, specifically, eyes with a 3-line decrease in BCVA.

### 10. ADMINISTRATIVE CONSIDERATIONS

# 10.1. Institutional Review Board (IRB) Approval

The IRB must review, approve, and provide continuing review of the clinical study protocol, protocol amendments, the informed consent documents, subject recruitment advertisements, and any other written information to be provided to the subjects. Initial IRB approval is an affirmative decision that the clinical study has been reviewed and may be conducted at the study site within the constraints set forth by the IRB, the institution, GCP, and applicable regulatory requirements. A copy of the IRB approval letter for the protocol, the informed consent, the intended advertising, and any written material to be provided to the subject must be submitted to Silk Technologies or designee prior to release of investigational supplies to the study site. Progress reports and notifications of serious adverse reactions will be provided to the IRB according to local regulations and guidelines. The IRB must be notified of completion or termination of the study. The study site must maintain an accurate and complete record of all reports, documents, and other submissions made to the IRB concerning this protocol.

## 10.2. Ethical Conduct of the Study

The study will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and in compliance with ICH guidelines, and all applicable US federal regulations and local legal and regulatory requirements.

# 10.3. Subject Information and Consent

A sample informed consent form containing the required elements of informed consent will be provided by Silk Technologies or designee. Any changes made to this sample must be approved by Silk Technologies or designee prior to submission to the IRB. After approval, the informed consent form must be submitted to and approved by the IRB. The informed consent must be written in a language in which the subject is fluent. Regulations require that foreign language informed consent forms be submitted to the IRB for approval. The foreign language translation is required to contain a statement of certification of the translation. The Investigator must forward a copy of the consent forms, the certified foreign language translation, and an IRB approval letter to Silk Technologies or designee.

It is the responsibility of the Investigator to inform each subject of the purpose of this clinical trial, including possible risks and benefits, and to document the informed consent process. Prior to undergoing any study-related procedures, the subject must read, sign, and date the current IRB-approved version of the informed consent form. The original informed consent form is to be retained by the study site, and a copy of the signed consent form is to be given to the subject.

# 10.4. Subject Confidentiality

Data generated for the study should be stored in a limited-access file area and be accessible only to representatives of the study site, Silk Technologies, the IRB, and FDA/relevant regulatory agencies. Medical information resulting from a subject's participation in this study

may be given to the subject's personal physician or to the appropriate medical personnel responsible for the subject's welfare. No information that can be related to a specific individual subject will be released or used in any fashion without the signed written consent of that subject. All reports and communications relating to study subjects will identify subjects only by initials and subject identification number. Complete subject identification will be kept by the Investigator for purposes of long-term follow-up, if needed. This information will be treated with strict adherence to professional standards of confidentiality.

## 10.5. Study Monitoring

The study will be monitored by Silk Technologies or designee in accordance with current GCP to assure compliance with the study protocol and the quality of the data collected. Monitoring visits will occur as required and could include a study initiation visit, monitoring visit(s), and a study close-out visit. Training will be provided for key investigative personnel in all aspects of study conduct. The Investigator will be responsible for making sure that site personnel are provided adequate training on conducting delegated tasks.

Before a site can enter a subject into the study, a representative of the Sponsor will:

- Determine the adequacy of the facilities
- Discuss with the Investigator(s) and other personnel their responsibilities regarding protocol adherence and the responsibilities of the Sponsor and or its representatives

This study will utilize eDC to optimize the eCRF source verification process. Monitors will review source data and overall study data/consistency remotely and onsite and query discrepancies based upon eCRF entries (eCRF initial entry is the source). During this monitoring, data are reviewed as entered by the site, and the monitors will flag any abnormalities, trends, or safety signals for Medical Monitor review and monitor follow-up onsite, if necessary. Refer to the Study Reference Manual and/or Regulatory Binder for details regarding data entry of study assessments and requirements for maintaining source documentation via paper/medical record.

During visits to the study site, the monitor may review the source documents including but not limited to signed informed consent forms, inclusion/exclusion checklist, medical/ocular history, concomitant medications, study assessments, study material accountability and storage, completed SANDE questionnaires and subject-completed VAS assessments, the reporting procedures for AEs, SAEs, and protocol deviations. The CRA will review the study documents maintained in the Regulatory Binder to ensure all documentation is current and only qualified and trained staff are appropriately delegated study related tasks. The CRA will also review the site-specific processes and research-related SOPs to ensure appropriate Investigator oversight is being maintained and documented as required by GCP/ICH.

All data generated during this study and the medical records/documents from which they originated are subject to inspection by the Sponsor or designee, the FDA, and other regulatory agencies. The Investigator must notify the Sponsor or designee promptly of any inspections scheduled by regulatory authorities.

Upon completion of the study, the clinical monitor will conduct a final visit (closeout) to the site. The objectives of this visit are to ascertain that all regulatory records and reports are complete, verify that the IP and other supplies have been accounted for (returned/destroyed), and ensure that the Investigators are aware of their responsibilities once the study ends.

The Investigator is responsible for permitting the Sponsor or designee direct access to any study documents for monitoring and auditing purposes, for providing adequate space for monitoring, and for addressing any questions or issues that might be raised by the monitor or auditor on a timely basis.

## 10.6. Case Report Forms and Study Records

The initial point of entry of study data should be the subject source documentation. The location and nature of the source documentation for all data collected in the study will be identified in the study files at the investigator's site.

Source document information should be legible. Recorded data should only be corrected by drawing a single line through the incorrect entry and writing the revision next to the corrected data. The person who has made the correction should place his or her initials as well as the date of the correction next to the correction. Data may not be obliterated by erasure, redaction, or with correction fluid.

Study data will be transcribed and recorded via an electronic data capture (EDC) system as electronic CRFs (eCRFs). Security and authorization procedures consistent with the EDC system must be used. At each subject visit, the appropriate eCRFs must be completed. Whenever an eCRF is used, be sure to provide all information requested including subject identification number, name or number of Investigator, date(s), etc. All applicable questions should be answered and all data requested should be provided. Those areas that require a response but are not filled in correctly are considered incomplete or erroneous entries, and will have to be corrected.

Each authorized study staff member will receive a unique access account in order to use the EDC system. Access accounts will not be shared among study staff. Authorized users will make entries and/or changes to eCRFs via a secure internet access. Each completed set of eCRFs will be reviewed by the Investigator who will then electronically sign and date the eCRF confirming that data for the subjects are complete and accurate.

The study records must include a copy of each Investigator's CV and medical license, completed, FDA Form 1572 or statement of Investigator, each eCRF, subject charts/source documents, Investigator's Brochure, protocol, protocol amendments, correspondence with the Sponsor and the IRB, IP storage, receipts, returns and dispensing records, Delegation Log, site training records, records of site monitoring, any unmasking documentation, AE and SAE reporting, IRB approvals, advertisements, written information provided to subjects, and subject completed ICFs. If the Investigator moves, withdraws from an investigation, or retires, the responsibility for maintaining the records may be transferred to another person (e.g., Sponsor, other Investigator) who will accept the responsibility. Notice of this transfer, including written acceptance, must be made to and agreed upon by the Sponsor.

#### 10.7. Protocol Deviations

The Investigator should not deviate from the requirements of this protocol except in the event of a medical emergency.

A reportable protocol deviation is defined as nonadherence to the protocol that involves inclusion/exclusion criteria, affects subject safety, or has the potential to affect the integrity of the data. All protocol deviations will be reported to Silk Technologies by entering the event in the appropriate eCRF page. Protocol deviations should be reported to the IRB in accordance with IRB-specific guidelines. If there is any question as to whether the deviation is reportable, Silk Technologies or designee and the IRB should be contacted.

All changes to the protocol will be made by the Sponsor or designee as an approved amendment to the protocol, submitted to the FDA, and approved by the IRB prior to implementation.

#### 10.8. Access to Source Documentation

A trial-related monitoring audit, review by the IRB, and/or regulatory inspection may be conducted at any time during or after completion of a study (Section 8). The Investigator will be given adequate notice if he/she is selected for an audit and must provide direct access to study documentation. The audit may include, but is not limited to, a review of all informed consent forms; a review of medical records; a review of regulatory documentation; an assessment of study conduct and protocol compliance; and a review of the study materials receipt, storage, and administration.

# 10.9. Data Generation and Analysis

Management of data and the production of the clinical study report will be the responsibility of Silk Technologies or its designee.

During the course of the trial, data queries will be generated for data items that are potentially erroneous and require appropriate clarification or correction. Such clarifications and corrections will be discussed with and approved by site personnel and appropriately documented. Prior to database lock, data listings will be generated, and anomalous values investigated.

#### 10.9.1. Retention of Data

Investigators should retain study-related records at the site until informed by the Sponsor. The Investigator will not move study documents or discard any records without notifying Silk Technologies. If the Principal Investigator moves from the current clinical site, Silk Technologies should be notified of the name of the person who will assume responsibility for maintenance of the records at the clinical site or the new address at which the records will be stored. The Investigator will notify Silk Technologies as soon as possible in the event of accidental loss or destruction of any study documentation. If it becomes necessary for Silk Technologies or designee, or the FDA or relevant regulatory authorities to review any documentation relating to the study, the Investigator must permit access to such records.

## 10.10. Publication and Disclosure Policy

All information concerning SDP-4 and the operations of Silk Technologies, such as patent applications, formulas, manufacturing processes, basic scientific data or formulation information not previously published, are considered CONFIDENTIAL and shall remain the sole property of Silk Technologies. The Investigator agrees to use this information only in accomplishing this study and will not use it for other purposes without the written consent of Silk Technologies

The publication policy is addressed in a separate agreement.

### 11. REFERENCE LIST

Abdel-Naby W, Cole B, Liu A, et al. Silk-Derived Protein Enhances Corneal Epithelial Migration, Adhesion, and Proliferation. Invest Ophthalmol Vis Sci. 2017;58(3):1425-33.

Craig JP, Nichols KK, Akpek EK, et al. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017;15:276-283.

Kim CE, Lee JH, Yeon YK, et al. Effects of silk fibroin in murine dry eye. Sci Rep. 2017;7:44364.

Lan W, Petnick A, Heryati S, et al. Nuclear factor kB: Central regulator in ocular surface inflammation and diseases. Ocul Surf. 2012;10:137-148.

Li N, Deng XG, He MF. Comparison of the Schirmer I test with and without topical anesthesia for diagnosing dry eye. Int J Ophthalmol. 2012;5:478-81.

Lemp MA. Report of the National Eye Institute/Industry workshop on Clinical Trials in Dry Eyes. CLAO J. 1995;21:221-32.

McMonnies CW, Chapman-Davies A. Assessment of conjunctival hyperemia in contact lens wearers. Part I. Am J Optom Physiol Opt. 1987;64:246-50. (McMonnies and Chapman-Davies, 1987a)

McMonnies CW, Chapman-Davies A. Assessment of conjunctival hyperemia in contact lens wearers. Part II. Am J Optom Physiol Opt. 1987;64:251-5. (McMonnies and Chapman-Davies, 1987b)

McMonnies CW, Ho A. Conjunctival hyperaemia in non-contact lens wearers. Acta Ophthalmol (Copenh). 1991;69:799-801.

Nichols KK, Mitchell GL, Zadnik K. The repeatability of clinical measurements of dry eye. Cornea. 2004;23:272-85.

Pflugfelder SC, Farley W, Luo L, et al. Matrix metalloproteinase-9 knockout confers resistance to corneal epithelial barrier disruption in experimental dry eye. Am J Ophthamol. 2005;166:61-71.

Smith VA, Rishmawi H, Hussein H, et al. Tear film MMP accumulation and corneal disease. Br J Ophthalmol. 2001;85:147-53.

Schaumberg DA, Gulati A, Mathers WD, et al. Development and validation of a short global dry eye symptom index. Ocul Surf. 2007;5:50-7.

Solomon A, Dursun D, Liu Z, et al. Pro- and anti-inflammatory forms of interleukin-1 in the tear fluid and conjunctiva of patients with dry eye disease. Invest Ophthalmol Vis Sci. 2001;42:2283-2292.

Tsubota K, Kaido M, Yagi Y, et al. Diseases associated with ocular surface abnormalities: the importance of reflex tearing. Br J Ophthalmol. 1999;83:89-91.

Wolffsohn JS, Arita R, Chalmers R, et al. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017;15:539-574.

### APPENDIX A. SPONSOR SIGNATURES

**Study Title:** 

A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-

Controlled, Parallel-Group, Study of SDP-4 Ophthalmic Solution in

Subjects with Dry Eye Disease (DED)

**Study Number:** 

SDP-4-CS202

**Final Date:** 

06 March 2020

This clinical study protocol was subject to critical review and has been approved by the Sponsor.

Signed:

Brian D. Lawrence, Ph.D.

Chief Executive Officer Silk Technologies, Ltd.

DocuSigned by:

Signed:

Brian Levy, O.D., M.Sc.

**Medical Monitor** 

Silk Technologies, Ltd.

Date: 12 Mar 2020

Date: 3/12/2020

# APPENDIX B. INVESTIGATOR'S SIGNATURE

| <b>Study Title:</b> | A Phase 2, Multicente<br>Controlled, Parallel-G<br>Subjects with Dry Eye | roup, Study of SDP-4 | ndomized, Vehicle-<br>Ophthalmic Solution in |
|---|---|---|---|
| <b>Study Number:</b> | SDP-4-CS202 | | |
| Final Date: | 06 March 2020 | | |
| Printed Name of Investigator | | | |
| Signature of Investigator | r | | |
| Date | | | |